CLINICAL TRIAL: NCT05087914
Title: Novel Non-opioid Post-surgical Pain Treatment in Females
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was not started, therefore recruitment did not happen
Sponsor: Northwestern University (Other)
Collaborators: Northwestern Medical Group (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Apkar Apkarian, Director Center for Translational Pain Research; Director Center of Excellence for Chronic Pain and Drug Abuse Research; Professor of Neuroscience; Anesthesia, and PM&R, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU00215128
Record Dates: First submitted 2021-10-11; First posted 2021-10-21 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Acute Pain; Bunionectomy; Toe Fusion
MeSH Terms: conditions — Acute Pain | interventions — carbidopa, levodopa drug combination; Naproxen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Carbidopa-Levodopa (100mg/25mg) + Naproxen (250mg) (Experimental): The study drug, Carbidopa-Levodopa, is an FDA-approved medicine traditionally used for the treatment of Parkinson's disease. The study drug will be used for an un-approved or un-labeled use: potentially managing pain in post-surgical patients. Carbidopa/Levodopa is an artificially made version of a naturally occurring hormone that helps regulate brain activity (Levodopa), combined with an artificially made version of a naturally occurring molecule that inhibits the breakdown of Levodopa (Carbidopa).
  Naproxen (250mg): Participants will receive one capsule TID, throughout the 5 days of the treatment period. Naproxen will be prescribed for active and control group.
  Interventions: Drug: Carbidopa-Levodopa (100mg/25mg):; Drug: Naproxen
- Placebo + Naproxen (250mg) (Placebo Comparator): Placebo:Participants will receive 1 the capsules on a three-times a day schedule for 5 days. A placebo looks like the study drug but is an inactive substance that has no medication. Researchers use a placebo to see if the study drug works better or is safer than not taking anything.
  Naproxen (250mg): Participants will receive one capsule TID, throughout the 5 days of the treatment period. Naproxen will be prescribed for active and control group.
  Interventions: Drug: Naproxen

INTERVENTIONS:
Drug: Carbidopa-Levodopa (100mg/25mg): — Participants will take 2 capsules (one containing naproxen, and the other containing either placebo or carbidopa/levodopa) 3 times per day (TID) for 5 days, the first dose is given right after the surgical procedure.
  Other Names: Sinemet; Parcopa; Rytary
  Arms: Carbidopa-Levodopa (100mg/25mg) + Naproxen (250mg)
Drug: Naproxen — Participants will take 2 capsules (one containing naproxen, and the other containing either placebo or carbidopa/levodopa) 3 times per day (TID) for 5 days, the first dose is given right after the surgical procedure.
  Other Names: Aleve; Anaprox; Naprosyn; Naprelan; Menstridol

SUMMARY:
This study aims to determine if treatment with Carbidopa/Levodopa and Naproxen in females (biological sex) with acute pain after a bunionectomy or toe fusion (24hrs, 48hrs and 5 days) will reduce pain when compared with females receiving Placebo and Naproxen.

DETAILED DESCRIPTION:
Acute post-surgical pain remains commonly treated with opioids. Although such treatments are efficacious, they can lead to opioid dependency. Disturbingly, opioid abuse often began as a direct consequence of prescription medications, primarily for pain management, and post-surgical pain management. Recent studies in from Apkarian lab suggest that the combination of dopamine and non-steroidal anti-inflammatory may be a safe, tolerable and efficacious novel post-surgical pain treatment option.

Therefore, the main hypothesis is: patients treated with Carbidopa/Levodopa and Naproxen will show a statistically significant decrease in post-surgical pain when compared with control intervention (Placebo plus Naproxen (250mg)). This will be done through a double-blind, randomized, placebo-controlled, parallel-group trial of the pharmacological treatment Carbidopa/Levodopa for females (N = 60) undergoing a bunionectomy or toe fusion surgery.

ELIGIBILITY:
Inclusion Criteria:

* female with no racial or ethnic restrictions;
* 18 to 75 years old;
* Have a bunionectomy or toe fusion surgery scheduled;
* must be able to read, understand, and sign consent form;
* generally healthy.

Exclusion Criteria:

* Chronic neurologic conditions, e.g., Parkinson's
* pregnancy;
* opioids use 60 mg/day oral morphine milligram equivalent.;
* use of anticoagulants (low dose ASA allowed);
* history of gastric ulcer; renal insufficiency or congestive heart failure,
* contraindication to study medication as determined by surgeon
* Any medical condition that in the investigator's judgment may prevent the individual from completing the study or put the individual at undue risk
* In the judgment of the investigator, unable or unwilling to follow protocol and instructions;
* Diagnosis of psychological diseases, such as major depression; bipolar disorder.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female (biological sex) with no racial or ethnic restrictions
Enrollment: 0 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Post-Surgical Pain using Numeric Rating Scale (NRS) | 1 and 4 weeks
  The primary endpoint will be the severity of pain measured by mean post surgical pain from surgery to end of intervention (~1 week) and end of the study, as indexed by a NRS. The NRS pain scale is a simple 10- point scale (0 = ''no pain'', 10 = ''pain as bad as you can imagine''). Mean pain during treatment will be compared between intervention groups.

SECONDARY OUTCOMES:
Patient Global Impression of Change (PGIC) | 1 and 4 weeks
  This questionnaire reflects a patient's belief about the efficacy of treatment. PGIC is a 7 point scale depicting a patient's rating of overall improvement. PGIC score will be compared between intervention groups.
Adverse Events | 1 and 4 weeks
  Participants will be query for possible adverse events during the intervention period (~1 weeks). Incidence of adverse events will be reported every visit.The frequency and severity of adverse effects will be compared between each intervention group.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF